CLINICAL TRIAL: NCT02052492
Title: A PHASE I, OPEN LABEL, DOSE-ESCALATION TRIAL EVALUATING THE SAFETY AND TOLERABILITY OF EF-022 (MODIFIED VITAMIN D BINDING PROTEIN MACROPHAGE ACTIVATOR) IN SUBJECTS WITH ADVANCED SOLID MALIGNANCIES
Brief Title: Safety Study of EF-022 ( Modified Vitamin D Binding Protein Macrophage Activator) in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Efranat Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR-001
Record Dates: First submitted 2014-01-30; First posted 2014-02-03 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Solid Tumors

ARMS (4):
- Cohort A: EF-022 100 ng once weekly (Experimental): Intra-Muscular injections of EF-022 100 ng once weekly for a period of 8 weeks
  Interventions: Drug: EF-022 (Modified Vitamin D Binding Protein Macrophage Activator)
- Cohort B: EF-022 500 ng once weekly (Experimental): Intra-Muscular injections of EF-022 500 ng once weekly for a period of 8 weeks
  Interventions: Drug: EF-022 (Modified Vitamin D Binding Protein Macrophage Activator)
- Cohort C: EF-022 1000 ng once weekly (Experimental): Intra-Muscular injections of EF-022 1000 ng once weekly for a period of 8 weeks
  Interventions: Drug: EF-022 (Modified Vitamin D Binding Protein Macrophage Activator)
- Expanded Cohort (Experimental): the expanded cohort, 24 Patients will be allocated to receive either 100ng, 500ng or 1000ng weekly treatment as detailed below: The first 18 patients will be assigned to alternating doses of either 100ng or 500ng in a sequential manner (each patient will be assigned to a single dose). A decision regarding adding a 1000ng dose cohort vs. continuing with the 100ng and 500ng doses will be based on a discussion of the interim analysis results.
  Interventions: Drug: EF-022 (Modified Vitamin D Binding Protein Macrophage Activator)

INTERVENTIONS:
Drug: EF-022 (Modified Vitamin D Binding Protein Macrophage Activator)

SUMMARY:
Activated macrophages, present in excess during natural inflammatory responses, bear the potential to kill and eradicate cancer cells. Macrophage activation has been demonstrated to require the serum-borne vitamin D binding protein (known as Gc protein), as well as B and T lymphocytes. However, in various cancer patients the Gc protein is deglycosylated by serum α-N-acetyl galactosaminidase (Nagalase) secreted from cancer cells. This deglycosylated Gc protein, lacking the N-acetylgalactosamine monosaccharide, cannot be converted to its form of Macrophage Activating Factor, leading to immunosuppression rather than Macrophage activation against cancer cells.

Efranat has developed cancer immunotherapy based on Macrophage Activating Factor produced from natural Gc protein extracted from FDA approved healthy human plasma.

In this phase I study, the treatment is given as Intramuscular, once-weekly injection of EF-022, for two courses, while each course is comprised of 4 injections.

The investigational treatment is expected to enhance immune response, thereby, improve patient's well being, quality of life and disease control.

Primary objectives:

1. To determine the safety and tolerability of EF-022 and to define the maximal tolerated dose (MTD) for potential administration.
2. To identify the Dose Limiting Toxicity (DLT) of EF-022.

Secondary objectives:

1. To determine the 'Recommended Phase 2 Dose' (RP2D) based on MTD data, immunological and pharmacodynamics markers
2. To explore preliminary efficacy of EF-022 in advanced solid tumors according to the 'Response Evaluation Criteria in the modified Solid Tumors' (RECIST 1.1) and blood levels of tumor-related markers known to reflect tumor burden.

Exploratory objectives:

1. To assess levels of immune-related factors in peripheral blood (determined by FACS analysis), reflecting induced immunological activities, including but not limited to, natural killer (NK), monocytes (M1 and M2) and T cell subpopulations (effector vs regulatory, CD4+ and CD8+ cells), B cells (CD20), myeloid and dendritic cells etc.
2. To assess the change in serum levels of protein biomarkers in the blood.
3. To immunohistochemically assess and compare tumor derived tissue samples Pre and post treatment. To analyze the infiltration of different population of cells into the tumor bed.

DETAILED DESCRIPTION:
Part 1:

Eligible subjects will be assigned, successively in order of accrual, to one of the three cohorts, to receive intramuscular (IM) injections of EF-022, once weekly for two courses of treatment. Each course will consist of 4 injections with one week intervals (total: 8 weeks of treatment).

Dose escalation will only proceed in the absence of dose-limiting toxicity (DLT) during course 1. For this purpose, each cohort will only begin its first course of EF-022 when the cohort preceding it has successfully completed its first 4-week treatment course without any signs of DLT. During this first course, should 1/3 patients experience DLT, dose escalation for the next cohort will not be authorized; the next cohort will receive the same dose as the one preceding it. If 2 patients or more of all patients treated with a given dose develop DLT, dose escalation will be halted and no more patients will be treated at the DLT dose. The value of MTD will be defined as the EF-022 dose below the dose at which DLT was seen for at least 2 subjects. Upon determination of the MTD, an additional cohort will be opened (confirmatory cohort) and treated with two courses of that dose.

Part 2:

During the expanded cohort, 24 Patients will be allocated to receive either 100ng, 500ng or 1000ng weekly treatment as detailed below: The first 18 patients will be assigned to alternating doses of either 100ng or 500ng in a sequential manner (each patient will be assigned to a single dose), with the caveat that given indications should be assigned equally, as much as possible, between these two doses.

Interim analysis will be performed once the 12th patient reaches Day 57 and the CT results as well as PD analysis are available for at least 12 patients, while at least 18 patients have begun study treatment. A decision regarding adding a 1000ng dose cohort vs. continuing with the 100ng and 500ng doses will be based on a discussion of the interim analysis results.

Each patient will receive 2 courses of treatment, i.e. weekly injections for a total period of 8 weeks, followed by a follow-up period of up to 12 months from the start of treatment (Day 1).

Continuation of treatment after the second course will be at the discretion of the investigator. Patients who will continue extended treatment post course 2 will keep the weekly injection dosage mode and continue therapy until disease progression, development of unacceptable toxicities, non-compliance, inter-current illness that prevents treatment continuation, withdrawal of consent, or change in subject condition that renders the subject unacceptable for further treatment.

All study patients who completed at least two courses of treatment will be followed up until 12 months from day 1 of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with inoperable, recurrent or metastatic tumor, deemed incurable, and who have either failed to respond to standard therapy or for whom no standard therapy is available or refuse to receive standard therapies or in case of SCC, the investigator decides that delay of the standard therapy does not have any risk for the patient.
2. Histologically or cytological-confirmed diagnosis of solid tumor on file. For the expanded cohort only the following immunological tumors will be recruited: epithelial ovarian cancer, cervical carcinoma, head & neck cancer, melanoma, kidney cancer (RCC), gastric cancer, lung cancer (SCLC or NSCLC), sarcoma, bladder cancer or squamous cell carcinoma (SCC) of the skin.
3. Measurable disease (i.e., present with at least one measurable lesion per modified RECIST, version 1.1).
4. Age: 18-80 years.
5. BMI: 18-36.
6. ECOG Performance Status 0 or 1.
7. Estimated life expectancy of at least 4 months.
8. Off prior chemotherapy, radiation therapy with curative intent, hormonal therapy, immunotherapy, biological therapies (excluded checkpoint inhibitors and Erbitux), immunosuppressive therapy [e.g., cyclosporine, humera, prograf, etc.] or immunomodulators [e.g., thalidomide, revlimid, etc.] for at least 4 weeks. Hormonal treatment is not allowed ONLY if given as an anti-cancer therapy. In any case the sponsor should be consulted prior to final decision.

   Prior treatment with checkpoint inhibitors (such as anti PD-1, anti PDL-1), and/or Erbitux, and/or palliative irradiation, does not require any wash out period before commencement of study drug treatment.

   Patients who were receiving mitomycin C, nitrosoureas, or carboplatin must be 6 weeks from the last administration of chemotherapy.
9. Patients must have adequate organ and marrow function within 7 days of first dosing. Hematology re-test results must keep meeting eligibility criteria on Day 1 of treatment prior to dosing.
10. All prior anti-cancer treatment-related toxicities (except alopecia and certain laboratory values) must be ≤ Grade 1 according to the Common Terminology Criteria for Adverse Events at the time of start of treatment. Stable grade 2 peripheral neuropathy secondary to neurotoxicity and/or chronic stable grade 2 radiotherapy related toxicity from prior therapies may be considered on a case by case basis.
11. No extensive radiotherapy (e.g., whole-pelvis, greater than 50% of neuroaxis, whole abdomen, whole body) within 12 months prior to start of study treatment.
12. No bone marrow transplantation within 3 years prior to start of study treatment.
13. Women and man of child bearing potential practicing an acceptable method of birth control during the study and at least 3 months after completion.
14. Female patient of childbearing potential has a negative serum pregnancy test within 7 days of first dose.
15. Understanding study procedures and willingness to comply for the entire length of the study and to provide written informed consent.
16. Patient has previously received maximum 3 regimens of systemic antineoplastic therapies.

Exclusion Criteria:

1. Current evidence of active and uncontrolled infection.
2. Known Cirrhosis.
3. Treatment refractory hypertension (blood pressure of systolic> 150 mmHg and/or diastolic > 95 mm Hg) which cannot be controlled by anti-hypertensive therapy;
4. A history or evidence of current Class IV congestive heart failure.
5. Current left ventricular ejection fraction < 50%
6. A history of acute coronary syndromes, coronary angioplasty.
7. Use of nonsteroidal anti-inflammatory drugs - including Aspirin - and/or any steroids within 7 days prior to start of study treatment (excluding eye drops and ointments). Those medications must be stopped or replaced by another equivalent permitted medication at least 7 days prior to Day 1. Those medications will be allowed within 7 days prior to start of treatment only if required as premedication prior to CT scan for patients who are allergic to the contrast media.
8. Patient has a known hypersensitivity to the components of study drug, its analogs, or drugs of similar chemical or biologic composition.
9. Patients with known brain metastases.
10. Patient has known psychiatric or substance abuse disorders that is uncontrolled and would interfere with cooperation with the requirements of the trial.
11. Patient is Human Immunodeficiency virus (HIV)-positive.
12. Evidence of active bleeding or bleeding diathesis, including blood or platelet transfusion within 14 days of the commencement of study treatment.
13. Patients with known chronic active hepatitis, hepatitis B virus (HBV) or hepatitis C virus (HCV) carriers.
14. Any known autoimmune disorders other than hypothyroidism or B12 deficiency.
15. Female subjects who are pregnant or nursing.
16. Use of alternative medicine (products only) and Herbal drugs with cancer treatment intent is not allowed within 7 days prior to start of study treatment and during the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-05; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events that meets the DLT definition | During first course of treatment (up to 4 weeks)
Percentage of participants with Adverse Events grade 3-4 | During two courses of treatment (up to 8 weeks)

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Rambam MC, Haifa
  - Sheba Medical Center, Ramat Gan